CLINICAL TRIAL: NCT06599736
Title: Effect of Temperature-Controlled Radiofrequency Ablation of the Posterior Nasal Nerve on Inflammatory Biomarkers in Patients With Allergic and Nonallergic Chronic Rhinitis
Brief Title: A Study of RhinAer Stylus for Treating Chronic Rhinitis
Acronym: BIOKLEAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aerin Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP1938
Record Dates: First submitted 2024-07-02; First posted 2024-09-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Rhinitis
Keywords: ENT; Chronic rhinitis; Allergic rhinitis; Non-allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic; Common Cold

STUDY DESIGN:
Intervention Model Description: Active treatment for all subject enrolling prospectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- RhinAer Stylus treatment (Experimental): The RhinAer procedure will be performed in the study clinic using the RhinAer Stylus and Aerin Console. The RhinAer Stylus is a disposable handheld device capable of delivering bipolar radiofrequency energy to tissue when connected to the Aerin Console radiofrequency generating device. Participants will have both nostrils treated in the portion of the nasal cavity mucosa overlying the region of the posterior nasal nerve.
  Interventions: Device: RhinAer Stylus

INTERVENTIONS:
Device: RhinAer Stylus — The RhinAer procedure incorporates use of the RhinAer Stylus (Model FG1393, CAT1394), which is a 510(k) cleared (FDA - K221907) disposable handheld device capable of delivering bipolar radiofrequency energy to tissue. The Aerin Console (Model FG226) RF generator with temperature control capable of delivering very low doses of energy is also cleared for use in the US (FDA - K162810).

SUMMARY:
Post-market study to continue to evaluate the effectiveness of the RhinAer Stylus for chronic rhinitis and the effect of treatment on inflammatory biomarkers.

DETAILED DESCRIPTION:
Prospective, Open Label, Multicenter Study of the Aerin Medical RhinAer® Stylus for Chronic Rhinitis to continue to evaluate the effectiveness of the RhinAer® Stylus for treating the posterior nasal nerve area to improve symptoms in adults diagnosed with chronic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 22 to 85 years (inclusively).
2. Willing and able to provide informed consent.
3. Willing and able to comply with the patient-specific requirements outlined in the study protocol.
4. Presenting to the ENT office seeking evaluation and/or treatment for chronic rhinitis (allergic or nonallergic) of at least 12 months duration
5. Willing to undergo the RhinAer procedure
6. Has a baseline rTNSS symptom score of ≥6 at time of screening
7. If on anticoagulation therapy, anticoagulant medications can be withheld during the perioperative period (at least 3-day window pre- and post-procedure).
8. Has been diagnosed with either allergic or non-allergic chronic rhinitis and meet the following criteria:

   * a. Allergic rhinitis: diagnosed with perennial (non-seasonal) allergic rhinitis and has demonstrated sensitization to specific allergens through skin prick testing, specific IgE blood testing, or other allergy testing methods, confirming the allergic nature of their rhinitis within the past 24 months.

OR

-b. Nonallergic rhinitis: diagnosed with nonallergic rhinitis with demonstration of a negative skin prick testing, specific IgE blood testing, or other allergy testing methods, confirming the nonallergic nature of their rhinitis within the past 24 months.

Exclusion Criteria:

1. Anatomic obstructions in the nasal passage(s) that in the investigator's opinion limits access to the posterior nasal nerve treatment area.
2. Has seasonal rhinitis symptoms.
3. Current or recent use of biologic therapy within past 3 months.
4. History of chronic epistaxis or has had episodes of significant nose bleeds in the past 3 months.
5. Known or suspected allergies or contraindications to the anesthetic agents and/or antibiotic medications to be used during the study procedure.
6. Known or suspected to be pregnant or is lactating.
7. Has any condition resulting in a predisposition to excessive bleeding (e.g., hereditary hemorrhagic telangiectasia [HHT]).
8. Has diagnosis of rhinitis medicamentosa, an active nasal or sinus infection or has a history of 'dry eye.'
9. Has had previous procedure or surgery for chronic rhinitis (e.g., PNN ablation).
10. Has had a nasal or sinus surgical procedure in the past six (6) months.
11. Currently participating in another clinical research study or has participated in an interventional study within the past 3 months.
12. Has a planned adjunctive procedure at the time of the study procedure or within the 6-month study follow-up period
13. Other medical conditions which in the opinion of the investigator would predispose the patient to poor wound healing, increased surgical risk, or poor compliance with the requirements of the study.

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in expression of nasal mucosal inflammatory markers in allergic and nonallergic chronic rhinitis patients | Baseline and 3 months post study procedure
  Change from baseline in expression of type-2 inflammatory cytokine markers in nasal mucus samples at 3 months post-procedure

SECONDARY OUTCOMES:
The change in cough and post-nasal drip symptoms | From baseline to 6 months post-procedure
  Change from baseline in cough and postnasal drip symptoms at 3 and 6 months post-procedure
The change in nasal symptoms of chronic rhinitis | From baseline to 6 months post-procedure
  Change from baseline in Reflective Total Nasal Symptom Score (rTNSS) total score at 3 and 6 months post-procedure. This is a 4 item questionnaire and each is scored from 0 (none) to 3 (severe), with a maximum score of 12. A higher number indicating more congestion.
Change in SNOT-22 score | From baseline to 6 months post-procedure
  Change from baseline in Sino-nasal Outcome Test (SNOT-22) score at 3 and 6 months post-procedure. The SNOT-22 contains 22 nose, sinus, and general health-related quality of life (HRQoL) items and is used to measure HRQoL associated with rhinosinusitis. Participants are required to indicate the level to which each listed nasal, sinus or HRQoL experience has been affected on a 6-point scale ranging from 0 (No problem) to 5 (Problem as bad as it can be).
Evaluate the impact of the RhinAer treatment in subjects with migraine-related symptoms | From baseline to 6 months post-procedure
  Change from baseline in Headache Impact Test (HIT-6) score at 3 and 6 months post-procedure. The HIT-6 is an instrument used to measure the adverse impact of headache on social functioning, role functioning, vitality, cognitive functioning and psychological distress as well as severity of headache pain. The HIT-6 requires patients to answer six questions regarding their migraines, each question is scored on a 5-point Likert scale.
  The HIT-6 scores range from 36 to 78. Higher scores indicate a greater impact of headaches on the respondent's life, i.e., Little or no impact (46 or less), Some impact (50 -55), Substantial impact (56-59) or Severe impact (60-78).
Evaluate medication usage in chronic rhinitis patients | From baseline to completion of study, an average of 6 months
  Change from baseline in medication usage at 3 months and 6 months post-procedure.
  Self-reported assessments of any change from baseline in frequency (including those taken as needed), dose, or change in route of administration of medications used to manage nasal symptoms related to chronic rhinitis, will be recorded. Assessment of medication use will be repeated at the time of procedure and at all subsequent follow-up timepoints, through completion of the study, an average of 6 months.
Evaluate patient reported pain outcomes related to the study procedure | Completed following the study procedure during treatment visit
  VAS will be completed by the patient immediately post-procedure.
  The Visual Analogue Scale (VAS) is a unidimensional measure of pain intensity that will be used to measure nasal pain associated with the procedure. A VAS is a 100-mm long horizontal line with verbal descriptors (word anchors) at each end to express the extremes of the feeling.
  Scores are obtained by measuring the distance in millimeters from the left origin of the line (0) to the point indicated with a slash placed by the patient to indicate their current level of pain in and around the nose. Results are then assigned a score between 0 and 100.

OTHER OUTCOMES:
Evaluate the occurrence of any device- or procedure-related adverse events | From baseline to completion of study, an average of 6 months
  Incidence, type, category, and severity of adverse events reported from time of consent through study completion, an average of 6 months.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Colorado ENT & Allergy, Colorado Springs, Colorado
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No
No data collected will be shared with other researchers participating in the study.